CLINICAL TRIAL: NCT06547996
Title: Effects of Transcranial Electrical Stimulation Combined With Retrieval Practice on Semantic Memory in Patients With Schizophrenia
Brief Title: Effects of tES Combined With Retrieval Practice on Semantic Memory in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast Normal University (Other)
Responsible Party: Principal Investigator, Xiaofeng Ma, Professor, Northeast Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.2023025
Record Dates: First submitted 2024-08-03; First posted 2024-08-12 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenic Patients

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS group (Experimental): In the tDCS group, the anode was placed over the left DLPFC (F3), and the cathode was placed over the contralateral supraorbital area (FP2). A direct current of 2mA was applied for 20 minutes during each stimulation session.
  Interventions: Device: tES-tDCS group
- tACS group (Experimental): In the tACS group, the anode was placed in the F3 region of the left dorsolateral prefrontal cortex (DLPFC), and the cathode was placed in the right supraorbital region (Fp2), and the current used was 2 mA AC at 40 Hz, with a stimulation time of 20 min.
  Interventions: Device: tES-tACS group
- sham group (Sham Comparator): In the sham group, the stimulation parameters, including the stimulation site and duration, were identical to those of the anodal group. However, during the 10-second ramp-up and ramp-down periods before and after stimulation, patients were unaware that the current was turned off.
  Interventions: Device: tES-sham group

INTERVENTIONS:
Device: tES-tDCS group — 2mA/20mins/session
  Arms: tDCS group
Device: tES-tACS group — 2mA/40Hz/20mins/session
  Arms: tACS group
Device: tES-sham group — 0mA/20mins/session
  Arms: sham group

SUMMARY:
The semantic processing deficit stands as a central feature of cognitive abnormalities in schizophrenia. Both transcranial electrical stimulation (tES) and retrieval practice have been demonstrated as external techniques capable of ameliorating the semantic processing deficit in individuals with schizophrenia. The inquiry examines whether the combined effect of tES and retrieval practice, following tES intervention targeting the left dorsolateral prefrontal cortex (L-DLPFC) in patients with schizophrenia, contributes to the preservation of semantic memory in these individuals.

Investigators plan to recruit 60 patients diagnosed with schizophrenia from hospitals. Treatment is administered by two examiners, each patient receives transcranial electrical stimulation（2mA×20min） with simultaneous learning of word lists. Each participant of each stimulation type was involved in both learning conditions, meaning that all participants completed both retrieval and restudy learning and testing Subsequently, Investigators observed their immediate and delayed memory performance through tests.

DETAILED DESCRIPTION:
1. Stimulation phase:

   In the tDCS group, the anode was placed over the left DLPFC (F3), and the cathode was placed over the contralateral supraorbital area (FP2). A direct current of 2mA was applied for 20 minutes during each stimulation session. In the tACS group, the anode was placed in the F3 region of the left dorsolateral prefrontal cortex (DLPFC), and the cathode was placed in the right supraorbital region (Fp2), and the current used was 2 mA AC at 40 Hz, with a stimulation time of 20 min. In the sham group, the stimulation parameters, including the stimulation site and duration, were identical to those of the anodal group. However, during the 10-second ramp-up and ramp-down periods before and after stimulation, patients were unaware that the current was turned off.
2. Learning phase:

   The experimental procedure followed the classic retrieval practice paradigm, which included a learning phase and a final test phase.

   During the experiment, participants were informed that they would learn two lists of words. Subsequently, they might either learn the words again or complete a list recall test, and will be given a final test shortly thereafter. The learning of the retrieval practice list and the restudy list was conducted in a randomly balanced manner. Each word was presented for 5 seconds, with a 500-millisecond interval between words. To avoid providing secondary retrieval cues between examples, all words were shuffled pseudo-randomly within categories. Each list contained 17 words, consisting of 5 examples from each of the 3 experimental categories (15 experimental examples, 2 filler examples). The first and last words presented in each list were filler words, thus controlling for the primacy and recency effects on memory.

   For the retrieval practice list, participants underwent two learning sessions and two retrieval sessions (S-T-S-T). During retrieval, participants were instructed to write down all the words they had just remembered within 5 minutes. For the restudy list, participants underwent four study sessions (S-S-S-S). Between each learning cycle, participants completed a 3-minute simple arithmetic task (dispersed attention task).
3. Testing phase:

Immediate Test: Participants were instructed to recall as many words as possible from the learned lists within 10 minutes after completing all learning tasks.

Delayed Test: Participants were informed to recall as many words as possible from the learned lists within 10 minutes 24 hours later.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5);
2. Aged 18 years or older, regardless of gender, with an educational level of elementary school or above;
3. All patients received stable-level antipsychotic medication treatment, were in a stable phase of disease treatment, able to understand the testing requirements, and cooperated to complete all research tasks;
4. No history of neurological disorders or other serious physical illnesses, and no history of intellectual disability;
5. No color blindness, color weakness, or other color vision impairments, with normal vision or corrected vision.

Exclusion Criteria:

1. Clear cognitive impairment caused by somatic or cerebral organic lesions, such as cerebrovascular diseases, traumatic brain injury, etc;
2. Individuals with mental disorders caused by substance dependence or abuse, or the use of psychoactive substances;
3. History of brain injury or other central nervous system-related organic diseases;
4. Individuals at significant risk of suicide or harming others;
5. Participation in similar experiments in the past 30 days prior to baseline.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
The correct recall rate of word lists | Immediate Test: 5minutes; Delayed Test: 24 hours
  The correct recall rate of word lists was calculated for each subject by the experimental assistant.
Adjusted Ratio of Clustering (ARC) | Immediate Test: 5minutes; Delayed Test: 24 hours
  Free recall organization was measured by the Adjusted Ratio of Clustering (ARC) scores. ARC scores range from 1 to 1. A 0 score indicates a level of clustering similar to what would be expected by chance, and a score of 1 implies perfect clustering. Negative values of ARC scores mean atypical and uninterpretable recall patterns. For that reason, negative scores were excluded from analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Ma, Professor, Principal Investigator — Northwest Normal University
Locations (1):
- Northwest Normal University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoy KE, Whitty D, Bailey N, Fitzgerald PB. Preliminary investigation of the effects of gamma-tACS on working memory in schizophrenia. J Neural Transm (Vienna). 2016 Oct;123(10):1205-12. doi: 10.1007/s00702-016-1554-1. Epub 2016 Apr 26. PMID 27116682
- [Background] Sreeraj VS, Shivakumar V, Sowmya S, Bose A, Nawani H, Narayanaswamy JC, Venkatasubramanian G. Online Theta Frequency Transcranial Alternating Current Stimulation for Cognitive Remediation in Schizophrenia: A Case Report and Review of Literature. J ECT. 2019 Jun;35(2):139-143. doi: 10.1097/YCT.0000000000000523. PMID 30024457
- [Background] Marko M, Cimrova B, Riecansky I. Neural theta oscillations support semantic memory retrieval. Sci Rep. 2019 Nov 27;9(1):17667. doi: 10.1038/s41598-019-53813-y. PMID 31776375
- [Background] Javadi AH, Cheng P. Transcranial direct current stimulation (tDCS) enhances reconsolidation of long-term memory. Brain Stimul. 2013 Jul;6(4):668-74. doi: 10.1016/j.brs.2012.10.007. Epub 2012 Oct 31. PMID 23137702
- [Background] Crossman M, Bartl G, Soerum R, Sandrini M. Effects of transcranial direct current stimulation over the posterior parietal cortex on episodic memory reconsolidation. Cortex. 2019 Dec;121:78-88. doi: 10.1016/j.cortex.2019.08.009. Epub 2019 Aug 28. PMID 31550617
- [Background] McKay AP, McKenna PJ, Bentham P, Mortimer AM, Holbery A, Hodges JR. Semantic memory is impaired in schizophrenia. Biol Psychiatry. 1996 Jun 1;39(11):929-37. doi: 10.1016/0006-3223(95)00250-2. PMID 9162204

DOCUMENTS (2):
  • Study Protocol (2024-08-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT06547996/Prot_000.pdf
  • Informed Consent Form (2024-08-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT06547996/ICF_001.pdf